CLINICAL TRIAL: NCT05743725
Title: Dexmedetomidine Versus Magnesium Sulphate in Patients Undergoing Craniotomy for Deeply Settled Intracranial Tumours
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ibraheem Abdelmageed, Dr.Ibraheem Abdelmageed, lecturer of anaesthesia and intensive care at Assiut university, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: master 2
Record Dates: First submitted 2022-11-26; First posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Brain Tumor
MeSH Terms: conditions — Brain Neoplasms | interventions — Dexmedetomidine; Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A: Dexmedetomidine (Active Comparator): Brain tumor excision under general anesthesia. This group will receive dexmedetomidine loading 1 microgram/kg bolus in 10 minutes followed by 0.2-1 microgram/kg/hour till the end of surgery.
  Interventions: Drug: Dexmedetomidine
- B: Magnesium sulphate (Active Comparator): Brain tumor excision under general anesthesia. This group will receive a 2 gm magnesium infusion for 30 minutes.
  Interventions: Drug: Magnesium sulfate

INTERVENTIONS:
Drug: Dexmedetomidine — dexmedetomidine loading 1 microgram/kg bolus in 10 minutes followed by 0.2-1 microgram/kg/hour till the end of surgery
  Arms: A: Dexmedetomidine
Drug: Magnesium sulfate — 2 gm magnesium infusion for 30 minutes
  Arms: B: Magnesium sulphate

SUMMARY:
An intracranial tumor, is an abnormal mass of tissue in which cells grow and multiply uncontrollably, seemingly unchecked by the mechanisms that control normal cells. More than 150 different brain tumors have been documented, but the two main groups of brain tumors are termed primary and metastatic.

Primary brain tumors include tumors that originate from the tissues of the brain or the brain's immediate surroundings.

Metastatic brain tumors include tumors that arise elsewhere in the body (such as the breast or lungs) and migrate to the brain, usually through the bloodstream Barbiturates, Thiopental and pentobarbital decrease CBF, cerebral blood volume (CBV), and ICP. The reduction in ICP with these drugs is related to the reduction in CBF and CBV coupled with metabolic depression. These drugs will also have these effects in patients who have impaired CO2 response.

Etomidate, as with barbiturates, etomidate reduces CBF, CMRo2, and ICP. Systemic hypotension occurs less frequently than with barbiturates. Prolonged use of etomidate may suppress the adrenocortical response to stress.

Dexmedetomidine as an anesthetic adjuvant improved hemodynamic stability and decreased anesthetic requirements in patients undergoing resection for brain tumors. In addition, DEX provided better surgical field exposure conditions and early recovery from anesthesia. Narcotics, in clinical doses, narcotics produce a minimal to moderate decrease in CBF and CMRo2. When ventilation is adequately maintained, narcotics probably have minimal effects on ICP. Despite its small ICP-elevating effect, fentanyl provides satisfactory analgesia and permits the use of lower concentrations of inhalational anaesthetics

DETAILED DESCRIPTION:
Anesthetic management:

Peripheral i.v line will be inserted and 2-3 mg midazolam is given. A pre-induction radial arterial line is inserted with the aid of infiltration of 2 ml lidocaine 2%. Invasive arterial blood pressure monitoring is started and pulse oximetry, 5-leads ECG, and NIBP are attached to the patient and mindray ipm-12 monitor is used. Anesthetic induction started with propofol 1-2 mg/kg, lidocaine 1 mg/kg, cis-atracurium 0.2 mg/kg and fentanyl 1-2 microgram/kg. Intubation is done with cuffed endotracheal tube and tidal volume and respiratory rate are set to achieve end-tidal Co2 of 30-28 mmHg. Esophageal temperature probe and urinary catheter are put in place. Patients then will receive maintenance of anesthesia with isoflurane < 1 MAC, propofol 10-60 microgram/kg/min, and cis-atracurium 2-3 microgram/kg/minute.

Patients are then grouped into two groups:

Group A: will receive dexmedetomidine loading 1 microgram/kg bolus in 10 minutes followed by 0.2-1 microgram/kg/hour till the end of surgery.

Group B: will receive 2 gm magnesium infusion for 30 minutes. All Patients will receive mannitol 20% 0.5-1 gm/kg and dexamethasone 8mg and paracetamol 1gm near the end of surgery. Patients will receive their fasting requirements of normal saline in the first 3 hours of surgery. Maintenance fluid used will be ringer acetate and will be given according to pulse pressure variation index (PPVI) that is derived from pulse contour analysis of invasive arterial blood pressure waveform. Patients will be given ringer acetate when PPVI is > 12%.

If hypotension occurred without change in PPVI targets, it will be treated with 10 mg ephedrine. On dural opening, brain relaxation score will be assessed which is a four points score 1. relaxed, 2. satisfactory, 3. firm, 4. Bulging. Arterial blood gas samples will be collected at induction and at the end of surgery. After removal of cranial fixation pins, anesthesia is discontinued and reversal of muscle relaxant is done with atropine 0.5 mg and neostigmine 0.05 mg/kg then extubation is done and patient is transferred to the ICU.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists (ASA) physical status I and II.
2. Age more than 18 years old.
3. supine Position
4. Patient undergoing craniotomy for deeply settled brain tumours.

Exclusion Criteria:

1. American Society of Anesthesiologists (ASA) physical status III or more and patients with GCS < 13
2. Other positions (prone position, lateral position)
3. Superficial brain tumors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-03-15 (Estimated); Primary Completion 2024-01-15 (Estimated); Study Completion 2024-02-15 (Estimated)

PRIMARY OUTCOMES:
Change in brain relaxation score | assessed by the neurosurgeon with dural opening, after 2 hours and before dural closure
  On dural opening, brain relaxation score will be assessed which is a four points score 1. relaxed, 2. satisfactory, 3. firm, 4. Bulging

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No